CLINICAL TRIAL: NCT02683525
Title: Phase II Trial of Inhibition of Dipeptidyl Peptidase (DPP)-4 With Sitagliptin for the Prevention of Acute Graft Versus-Host Disease Following Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Sitagliptin for Prevention of Acute Graft Versus-Host Disease After Allogeneic Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sherif S. Farag (Other)
Responsible Party: Sponsor-Investigator, Sherif S. Farag, Lawrence H. Einhorn Professor of Oncology, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUSCC-0522
Record Dates: First submitted 2016-02-02; First posted 2016-02-17 (Estimated); Results first posted 2020-12-29 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Graft vs Host Disease; Hematopoietic Stem Cell Transplantation
Keywords: Allogeneic; Sitagliptin
MeSH Terms: conditions — Graft vs Host Disease | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sitagliptin (Experimental): Sitagliptin 600 mg q 12 hours PO starting on Day -1 before transplant to be administered between 8:00 am and 10:00 am then given every 12 hours (total 32 doses) through day +14.
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — 600 mg ever 12 hours by mouth will be given starting the day before transplant through day +14 after transplant

SUMMARY:
Primary Objective

Evaluate the efficacy of sitagliptin in reducing the incidence of grade II-IV acute Graft Versus-Host Disease (GvHD) by day +100 post-transplant in patients undergoing allogeneic hematopoietic stem cell transplantation and receiving standard sirolimus and tacrolimus GvHD prophylaxis.

Secondary Objectives

The following descriptive secondary objectives will be studied:

1. Describe the tolerability and potential toxicity of sitagliptin.
2. Describe the cumulative incidence of grades II-IV acute GvHD by day +100.
3. Describe the cumulative incidence of grades III-IV acute GvHD.
4. Describe the engraftment kinetics of absolute neutrophil count and platelets.
5. Describe the incidence of infections occurring during the 100 days post-transplant.
6. Describe non-relapse mortality (NRM) at day +30, +100, and 1 year post-transplant.
7. Describe overall survival.
8. Describe the incidence of chronic GvHD.
9. Describe the cumulative incidence of relapse of the primary hematological malignancy.

DETAILED DESCRIPTION:
This is an open label phase II study in patients undergoing allogeneic hematopoietic stem cell transplantation and receiving standard sirolimus and tacrolimus GvHD prophylaxis. Although the myeloablative preparative regimen is not prescribed, it is anticipated that most patients will receive total body irradiation (TBI) plus etoposide (TBI/VP16), or high-dose thiotepa plus cyclophosphamide according to institutional standards. Regardless of the preparative regimen, all patients will receive the following regimen for GvHD prophylaxis, which includes the study drug sitagliptin:

Day -3: Tacrolimus is initiated on day -3 with a suggested starting dose of 0.01 mg/kg/day IV as a continuous infusion and them modified to target a serum level of 5-10 ng/ml. Serum levels should be monitored at least twice weekly until discharge, then at times of outpatient clinic visits according to institutional practice. Tacrolimus may be switched to PO dosing when the patient is able to tolerate oral intake satisfactorily. Note that concurrent use of agents such as itraconazole, voriconazole or fluconazole (at doses > 200 mg) may inhibit the metabolism of tacrolimus, and thus increase tacrolimus levels. Initial dosing may be decreased in order to account for increased levels related to use of 'azole' agents. In addition, it is recommended to check tacrolimus levels twice weekly when these agents are initiated concurrently.

Sirolimus is started on day -3 with a suggested loading dose of 1 mg PO, then 0.5 mg/day PO single dose from day -2 to maintain a target serum level of 5-10 ng/ml. Serum levels should be monitored twice weekly until discharge, then at times of outpatient clinic visits according to institutional practice. Initial dosing may be decreased in order to account for increased levels related to use of 'azole' agents.

Day -1: Sitagliptin 600 mg q 12 hours PO starting on Day -1 to be administered between 8:00 am and 10:00 am then given every 12 hours (total 32 doses) through day +14.

In the absence of acute GvHD, begin tapering of both tacrolimus and sirolimus on Day +100 as tolerated with a goal of stopping by Day +180. The rate of taper may be adjusted for presence of signs and symptoms of GvHD. Mycophenolate mofetil may be substituted for tacrolimus or sirolimus if any toxicity related to these drugs arises (e.g., renal failure, hemolytic microangiopathy, allergic rash, etc.).

ELIGIBILITY:
INCLUSION CRITERIA:

A. Patients with any of the following hematologic malignancies:

1. Acute myeloid leukemia (AML) with any of the following:

   1. In first remission (CR1) with intermediate risk or high-risk cytogenetic and/or molecular features.
   2. Patients in second or subsequent complete remission (CR2, CR3, etc.).
   3. Primary refractory or relapsed AML with no more than any one of the following adverse additional features according to modified CIBMTR criteria:49

      * Duration of first CR < 6 months
      * Poor risk cytogenetics or molecular features (FLT-3 internal tandem duplication (ITD); complex karyotype with ≥3 clonal abnormalities, 5q-/-5, 7q-/-7, 11q23 abnormalities, inv(3), monosomal karyotype)
      * Circulating peripheral blood blasts at time of enrollment
      * Karnofsky performance status <90%
2. Acute lymphoblastic leukemia (ALL) with any of the following:

   1. In CR1 or subsequent complete remission (CR2, CR3, etc.)
   2. Primary refractory or relapsed ALL with no more than one of the following adverse features according to modified CIBMTR criteria:49

      * Second or subsequent relapse
      * Bone marrow blasts >25% at time of enrollment
      * Age >40 years
3. Myelodysplasia with any of the following features:

   1. Refractory anemia with excess blasts type I (5-10% blasts) or II (11-20% blasts) in the bone marrow (RAEB I and II)
   2. Refractory cytopenia with multilineage dysplasia (RCMD) and poor risk cytogenetics (i.e., chromosome 7 abnormalities or complex karyotype with at least 3 abnormalities per clone)
4. Chronic myelogenous leukemia (CML) with one of the following criteria:

   1. Accelerated phase, defined by any of the following:

      * Blasts 10-19% in peripheral blood white cells or bone marrow
      * Peripheral blood basophils at least 20%
      * Persistent thrombocytopenia (<100 x 109/l) unrelated to therapy, or persistent thrombocytosis (>1000 x 109/l) unresponsive to therapy
      * Increasing spleen size and increasing white blood cell (WBC) count unresponsive to therapy
      * Cytogenetic evidence of clonal evolution (i.e., the appearance of an additional genetic abnormality that was not present in the initial specimen at the time of diagnosis of chronic phase)
   2. Chronic phase provided a complete hematologic remission was not achieved by 3 months or a complete cytogenetic remission by 18 months and the patient had received at least 2 tyrosine kinase inhibitors
5. Patients with aggressive non-Hodgkin's lymphoma (NHL), including diffuse large cell lymphoma, mediastinal B-cell lymphoma, transformed lymphoma, mantle cell lymphoma, and peripheral T cell lymphoma, who also have one of the following criteria:

   1. Failure to achieve complete remission to primary induction therapy
   2. Relapsed and refractory to at least one line of salvage systemic therapy
   3. Failed stem cell collection
6. Patients with Hodgkin's lymphoma meeting one of the following criteria:

   1. Primary refractory (failure to achieve complete remission to primary induction therapy)
   2. Relapsed and refractory to at least one line of salvage systemic therapy
   3. Failed stem cell collection

B. Patient age ≥ 18 to ≤ 60 years

C. Karnofsky Performance status ≥ 70%

D. Patients must also receive a full myeloablative preparative regimen (Patients treated with either total body irradiation (TBI)-based or high-dose chemotherapy only regimens are eligible other than high-dose busulfan containing regimens or regimens that include anti-thymocyte globulin or other T cell depleting antibodies)

E. Patients receiving allogeneic peripheral blood stem cell (PBSC) grafts from HLA-matched (5/6 and 6/6 matches) siblings or from well matched unrelated donors (9/10 or 10/10 matches at HLA-A, B, C, DRB1 and DQB1 by high resolution typing) are included. All grafts will be unmanipulated (i.e., no T cell depleted or CD34 selected grafts).

F. No uncontrolled bacterial, viral or fungal infection at time of enrollment defined as currently taking medication and progression of clinical symptoms

G. No HIV disease (Patients with immune dysfunction are at a significantly higher risk of infection from intensive immunosuppressive therapies)

H. Non-pregnant and non-nursing

I. Required baseline values within 60 days prior to admission:

1. LVEF ≥ 45%
2. DLCO ≥ 50% of predicted (corrected for hemoglobin)

J. Required baseline laboratory values within 16 days prior to admission:

1. Estimated creatinine clearance ≥60 ml/min
2. Serum total bilirubin ≤ 2 x upper limit of normal value (ULN)
3. AST and ALT ≤ 2 x ULN (unless determined by treating physician to be related to underlying malignancy)

K. Signed written informed consent (Patient must be capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent)

L. Patients must otherwise fulfill institutional criteria for eligibility to undergo myeloablative allogeneic stem cell transplantation

EXCLUSION CRITERIA:

A. Symptomatic uncontrolled coronary artery disease or congestive heart failure

B. Severe hypoxemia with room air PaO2 < 70, supplemental oxygen dependence, or DLCO < 50% predicted

C. Patients with active central nervous system involvement

D. Prior allogeneic or autologous hematopoietic stem cell transplant in past 12 months

E. Patients with diabetes mellitus requiring insulin secretagogues and/or insulin

F. Patients with hypertriglyceridemia with serum triglyceride level ≥500 mg/d (lipid lowering drugs may be used to control level)

G. Patients with a history of pancreatitis

H. Patients with symptomatic cholelithiasis

I. Patients with a current dependence on alcohol (characterized by a physical addiction to alcohol that interferes with physical or mental health, and social, family or job responsibilities)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Farag, MD, PhD, Principal Investigator — Indiana University School of Medicine, Indiana University Simon Cancer Center
Locations (2):
- United States (2):
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana

REFERENCES:
- [Derived] Farag SS, Abu Zaid M, Schwartz JE, Thakrar TC, Blakley AJ, Abonour R, Robertson MJ, Broxmeyer HE, Zhang S. Dipeptidyl Peptidase 4 Inhibition for Prophylaxis of Acute Graft-versus-Host Disease. N Engl J Med. 2021 Jan 7;384(1):11-19. doi: 10.1056/NEJMoa2027372. PMID 33406328

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sitagliptin
Started | 37
Completed | 29
Not Completed | 8
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1
Not completed — Disease Progression | 6

BASELINE CHARACTERISTICS:
Arm/Group | Sitagliptin
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (10.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 35
  More than one race | 0
  Unknown or Not Reported | 1
Disease Type [Count of Participants; unit: Participants]
  Acute Lymphoblastic Leukemia (ALL) | 9
  Acute Myeloid Leukemia (AML) | 20
  Chronic Myeloid Leukemia (CML) | 4
  Myelodysplasia (MDS) | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Grade II-IV Acute GvHD by Day +100 Following Transplant
Description: Percent of patients and the 95% Confidence interval who did not have Grade II-IV Acute GvHD by 100 days following transplant. Since the study completed the two-phase design, proper inference was used to generate the confidence interval (Koyama and Chen). Only patients who were on the study for at least 100 days post transplant were included in the analysis.
Time Frame: up to 100 days
Population: Patients on study at least 100 days post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sitagliptin
Number analyzed (Participants) | 36
percentage of participants | 94.4 [82.0 to 97.1]

2. Secondary Outcome: Percentage of Patients With Grade II-IV Acute GvHD at Day +100
Description: Kaplan-Meier methods will be used to conduct a competing risk analysis. Time until grade II-IV acute GvHD will be calculated from transplant until grade II-IV acute GvHD or death from GvHD. Patients who relapsed or died from causes other than GvHD will be considered a competing risk and calculated from time of transplant until relapse or death. Otherwise, patients will be censored and calculated from transplant until the last known alive date. The cumulative incidence percentage of grade II-IV acute GvHD at day +100 was calculated along with a 95% confidence interval.
Time Frame: 100 days from transplant
Population: All patients who received a transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sitagliptin
Number analyzed (Participants) | 37
percentage of participants | 5.5 [1.0 to 16.3]

3. Secondary Outcome: Number of Patients With Treatment Related Adverse Events Grade 3 or Higher for Non-hematological Toxicity
Description: Number of unique patients who had a treatment related (possible, probable or definite) non-hematological adverse event that was graded 3 or greater.
Time Frame: up to 2 months
Population: All patients who received a transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin
Number analyzed (Participants) | 37
Participants | 0

4. Secondary Outcome: Percentage of Patients With Grade III-IV Acute GvHD at Day +100
Description: Kaplan-Meier methods will be used to conduct a competing risk analysis. Time until grade III-IV acute GvHD will be calculated from transplant until grade III-IV acute GvHD or death from GvHD. Patients who relapsed or died from causes other than GvHD will be considered a competing risk and calculated from time of transplant until relapse or death. Otherwise, patients will be censored and calculated from transplant until the last known alive date. The cumulative incidence percentage of grade II-IV acute GvHD at day +100 was calculated along with a 95% confidence interval.
Time Frame: 100 days from transplant
Population: All patients who received a transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sitagliptin
Number analyzed (Participants) | 37
percentage of participants | 2.7 [0.2 to 12.3]

5. Secondary Outcome: Median Time to Engraftment of Neutrophils
Description: Time to neutrophil engraftment will be analyzed by the Kaplan-Meier method. The time to engraftment of neutrophils is defined as the time from day 0 to the date of the first of three consecutive days after transplantation during which the absolute neutrophils count (ANC) is at least 0.5 x109/l. Patients who did not have neutrophil engraftment before death will be censored at the date of death. The median and 95% confidence intervals were calculated.
Time Frame: up to 1 month
Population: All patients who received a transplant
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sitagliptin
Number analyzed (Participants) | 37
days | 13 [12 to 15]

6. Secondary Outcome: Median Time to Engraftment of Platelets
Description: Time to platelet engraftment will be analyzed by the Kaplan-Meier method. The time to engraftment of platelets is defined as the time from day 0 to the first of seven consecutive Complete Blood Counts (CBCs) obtained on different days after transplantation during which the platelet count is at least 20 x109/l. The CBCs obtained should be at least seven days after the most recent platelet transfusion. The median and 95% confidence intervals were calculated.
Time Frame: up to 4 months
Population: All patients who received a transplant.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sitagliptin
Number analyzed (Participants) | 37
days | 15 [14 to 16]

7. Secondary Outcome: Number of Unique Patients With Infections by Day +100
Description: Number of unique patients who had each type of infection (i.e., viral, bacterial, fungal, etc.) during the 100 days post transplant. A patient could have more than one type of infection.
Time Frame: 100 days from transplant
Population: All patients who received a transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin
Number analyzed (Participants) | 37
Participants
  Bacterial | 5
  Gram Positive Bacteria | 1
  Other Bacteria | 1
  Fungal | 1
  Viral | 11
  CMV | 1

8. Secondary Outcome: Percentage of Patients With Non-relapse Mortality (NRM) at +1 Year
Description: Kaplan-Meier methods will be used to conduct a competing risk analysis. Time until non-relapse death will be calculated from transplant until death. Patients who died from relapse will be considered a competing risk and calculated from time of transplant until death. Otherwise, patients will be censored and calculated from transplant until the last known alive date. The cumulative incidence percentage of non-relapse mortality at day +365 was calculated along with a 95% confidence interval.
Time Frame: 1 year from transplant
Population: All patients who received a transplant.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sitagliptin
Number analyzed (Participants) | 37
percentage of participants | 0 [NA to NA] — Since no patients died from non-relapse mortality by 1 year, a confidence interval was not generated.

9. Secondary Outcome: Percentage of Patients Surviving at +1 Year
Description: Duration of time from the start of treatment to time of death due to any causes. Patients who do not die will be censored on their last known alive date. Kaplan-Meier methods will be used and the median and 95% confidence intervals will be calculated. The cumulative incidence percentage of survival at day +365 was calculated along with a 95% confidence interval.
Time Frame: 1 year from transplant
Population: All patients who received a transplant.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sitagliptin
Number analyzed (Participants) | 37
percentage of participants | 94.3 [79.0 to 98.5]

10. Secondary Outcome: Percentage of Patients Diagnosed With Chronic GvHD at 1 Year
Description: Patients surviving at least 100 days will be evaluable for chronic GvHD. The cumulative incidence of chronic GvHD (total, and mild, moderate, severe) will be described using deaths from causes other than chronic GvHD considered as a competing risk. Kaplan-Meier methods will be used to conduct a competing risk analysis. Time until chronic GvHD will be calculated from transplant until chronic GvHD or death from GvHD. Patients who relapsed or died from causes other than GvHD will be considered a competing risk and calculated from time of transplant until relapse or death. Otherwise, patients will be censored and calculated from transplant until the last known alive date. The cumulative incidence percentage at 1 year will calculated along with a 95% confidence interval.
Time Frame: 1 year from transplant
Population: Patients on study at least 100 days post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sitagliptin
Number analyzed (Participants) | 36
percentage of participants | 37.4 [21.5 to 53.4]

11. Secondary Outcome: Percentage of Patients With Relapse of the Primary Hematological Malignancy at 1 Year
Description: Kaplan-Meier methods will be used to conduct a competing risk analysis. Time until relapse will be calculated from transplant until relapse or death from relapse. Patients who died from causes other than relapse will be considered a competing risk and calculated from time of transplant until death. Otherwise, patients will be censored and calculated from transplant until the last known alive date. The cumulative incidence percentage of relapse at day +365 was calculated along with a 95% confidence interval.
Time Frame: 1 year from transplant
Population: All patients who received a transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sitagliptin
Number analyzed (Participants) | 37
percentage of participants | 25.6 [12.5 to 40.9]

ADVERSE EVENTS:
Time Frame: Up to 2 months for Adverse Events (Serious and Other). Up to 2 years for all cause mortality.
Arm/Group | Sitagliptin
All-Cause Mortality (participants affected / at risk) | 4/37
Serious Adverse Events (participants affected / at risk) | 6/37
Other Adverse Events (participants affected / at risk) | 32/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=37)
Multi-organ failure (General disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=37)
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Hemolysis (Blood and lymphatic system disorders) | 2
Diarrhea (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 22
Edema limbs (General disorders) | 2
Bladder infection (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Anorexia (Metabolism and nutrition disorders) | 10
Headache (Nervous system disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT02683525/Prot_SAP_000.pdf